CLINICAL TRIAL: NCT01874691
Title: China Acute Myocardial Infarction Registry
Acronym: CAMIRegistry
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yuejin Yang, Doctor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2011BAI11B02-A; 2011BAI11B02 (Other Grant/Funding Number: Chinese Ministry of Science and Technology)
Record Dates: First submitted 2013-06-04; First posted 2013-06-11 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; China; Registry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute myocardial infarction: acute myocardial infarction including ST-elevation and non ST-elevation myocardial infarction

SUMMARY:
This study is to build a Chinese national registry and surveillance system for acute myocardial infarction(AMI) to obtain real-world information about current status of characteristics, risk factors, diagnosis, treatment and outcomes of Chinese AMI patients; And to propose scientific precaution strategies aimed to prevent effectively from the incidence of AMI; And to optimize the management and outcomes of AMI patients through implementation of guideline recommendations in clinical practice, and analysis and development of effective treatment strategies; And to create cost-effective assessment system.

DETAILED DESCRIPTION:
The aim of the study is to establish the national platform for surveillance, clinical research and translational medicine in China, designed to facilitate efforts to improve the quality of AMI patient care and thus decrease morbidity and mortality associated with AMI.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must be admitted within 7 days of acute ischemic symptoms and diagnosed acute ST-elevation or non ST-elevation myocardial infarction. Diagnosis criteria must meet Universal Definition for AMI (2012). All participating hospitals are required to enroll consecutive patients with AMI.

Exclusion Criteria:

* Myocardial infarction related to percutaneous coronary intervention and coronary artery bypass grafting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients admitted within 7 days of acute ischemic symptoms and diagnosed acute ST-elevation or non ST-elevation myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality of the patients with acute myocardial infarction in different-level hospitals across China | the duration of hospital stay, an expected average of 2 weeks
  Different-level hospitals include Provincial-level, city-level, County-level hospitals from all over China.

SECONDARY OUTCOMES:
The rate of the application of thrombolysis and primary percutaneous coronary intervention for Chinese patients with acute myocardial infarction in different-level hospitals | 24 hours
  In different-level hospitals, How many patients with acute myocardial infarction receive thrombolysis and/or primary percutaneous coronary intervention within 24 hours from the onset,respectively?
provoking factors of Chinese patients with AMI across different areas and different population in China | 24 hours
  The different factors that can provoke the onset of acute myocardial infarction, for example, excess exercise, overload work, heavy smoking, heavy drinking of alcohol and so on.

OTHER OUTCOMES:
the in-hospital cost of Chinese patients with acute myocardial infarction | the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, MD., Study Chair — Fuwai Hospital, Chinse Academy of Medical Sciences
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Peterson ED, Roe MT, Rumsfeld JS, Shaw RE, Brindis RG, Fonarow GC, Cannon CP. A call to ACTION (acute coronary treatment and intervention outcomes network): a national effort to promote timely clinical feedback and support continuous quality improvement for acute myocardial infarction. Circ Cardiovasc Qual Outcomes. 2009 Sep;2(5):491-9. doi: 10.1161/CIRCOUTCOMES.108.847145. PMID 20031882
- [Derived] Song Z, Danzeng C, Jiang Y, Yang J, Yang W, Qian H, Yang Y. Association Between Admission Blood Pressure and In-hospital Mortality and Long-term Mortality of Patients With ST-elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention: A China Acute Myocardial Infarction Registry Study. Rev Cardiovasc Med. 2025 Aug 30;26(8):33512. doi: 10.31083/RCM33512. eCollection 2025 Aug. PMID 40927077
- [Derived] Wu C, Zhang Z, Su S, Xu H, Song L, Wu Y, Qiao S, Wang Y, Li W, Tang Y, Gao X, Yang J, Yang Y; China Acute Myocardial Infarction Registry Study Group. Role of heavy sweating for ST-segment elevation myocardial infarction: analysis of the China Acute Myocardial Infarction registry. BMC Cardiovasc Disord. 2025 May 20;25(1):385. doi: 10.1186/s12872-025-04840-3. PMID 40394465
- [Derived] Yang J, Li Y, Li X, Tao S, Zhang Y, Chen T, Xie G, Xu H, Gao X, Yang Y. A Machine Learning Model for Predicting In-Hospital Mortality in Chinese Patients With ST-Segment Elevation Myocardial Infarction: Findings From the China Myocardial Infarction Registry. J Med Internet Res. 2024 Jul 30;26:e50067. doi: 10.2196/50067. PMID 39079111
- [Derived] Xu X, Wang Z, Yang J, Fan X, Yang Y. Burden of cardiac arrhythmias in patients with acute myocardial infarction and their impact on hospitalization outcomes: insights from China acute myocardial infarction (CAMI) registry. BMC Cardiovasc Disord. 2024 Apr 23;24(1):218. doi: 10.1186/s12872-024-03889-w. PMID 38654151
- [Derived] Yang J, Zhao Y, Wang J, Ma L, Xu H, Leng W, Wang Y, Wang Y, Wang Z, Gao X, Yang Y; China Acute Myocardial Infarction Registry Research Group. Current status of emergency medical service use in ST-segment elevation myocardial infarction in China: Findings from China Acute Myocardial Infarction (CAMI) Registry. Int J Cardiol. 2024 Jul 1;406:132040. doi: 10.1016/j.ijcard.2024.132040. Epub 2024 Apr 16. PMID 38614365
- [Derived] Jiang Y, Yang JG, Qian HY, Yang YJ. Association between living alone and all-cause mortality of young and middle-aged patients with acute myocardial infarction: analysis of the China Acute Myocardial Infarction (CAMI) registry. BMC Public Health. 2024 Jan 2;24(1):14. doi: 10.1186/s12889-023-17486-7. PMID 38166780
- [Derived] Wu C, Gao X, Li L, Jing Q, Li W, Xu H, Zhang W, Li S, Zhao Y, Wang Y, Li W, Wu Y, Hu F, Jin C, Qiao S, Yang J, Yang Y; CAMI (China Acute Myocardial Infarction) Registry Study Group. Role of ST-Segment Resolution Alone and in Combination With TIMI Flow After Primary Percutaneous Coronary Intervention for ST-Segment-Elevation Myocardial Infarction. J Am Heart Assoc. 2023 Jul 18;12(14):e029670. doi: 10.1161/JAHA.123.029670. Epub 2023 Jul 14. PMID 37449560
- [Derived] Cui K, Fu R, Yang J, Xu H, Yin D, Song W, Wang H, Zhu C, Feng L, Wang Z, Wang Q, Lu Y, Dou K, Yang Y; CAMI Registry Investigators. The impact of fasting stress hyperglycemia ratio, fasting plasma glucose and hemoglobin A1c on in-hospital mortality in patients with and without diabetes: findings from the China acute myocardial infarction registry. Cardiovasc Diabetol. 2023 Jul 4;22(1):165. doi: 10.1186/s12933-023-01868-7. PMID 37403082
- [Derived] Lv J, Wang C, Gao X, Yang J, Zhang X, Ye Y, Dong Q, Fu R, Sun H, Yan X, Zhao Y, Wang Y, Xu H, Yang Y; China Acute Myocardial Infarction Registry study group. Development and validation of dynamic models to predict postdischarge mortality risk in patients with acute myocardial infarction: results from China Acute Myocardial Infarction Registry. BMJ Open. 2023 Mar 29;13(3):e069505. doi: 10.1136/bmjopen-2022-069505. PMID 36990493
- [Derived] Zhao X, Wang J, Yang J, Chen T, Song Y, Li X, Xie G, Gao X, Xu H, Gao R, Yuan J, Yang Y. Machine learning for prediction of bleeding in acute myocardial infarction patients after percutaneous coronary intervention. Ther Adv Chronic Dis. 2023 Mar 4;14:20406223231158561. doi: 10.1177/20406223231158561. eCollection 2023. PMID 36895330
- [Derived] Wu C, Li L, Wang S, Zeng J, Yang J, Xu H, Zhao Y, Wang Y, Li W, Jin C, Gao X, Yang Y, Qiao S. Fibrinolytic therapy use for ST-segment elevation myocardial infarction and long-term outcomes in China: 2-year results from the China Acute Myocardial Infarction Registry. BMC Cardiovasc Disord. 2023 Feb 22;23(1):103. doi: 10.1186/s12872-023-03105-1. PMID 36814182
- [Derived] Fu R, Cui K, Yang J, Xu H, Yin D, Song W, Wang H, Zhu C, Feng L, Wang Z, Wang Q, Lu Y, Dou K, Yang Y; CAMI Registry Investigators. Fasting stress hyperglycemia ratio and in-hospital mortality after acute myocardial infarction in patients with different glucose metabolism status: Results from China acute myocardial infarction registry. Diabetes Res Clin Pract. 2023 Feb;196:110241. doi: 10.1016/j.diabres.2023.110241. Epub 2023 Jan 6. PMID 36623641
- [Derived] Wei ZY, Yang JG, Qian HY, Yang YJ; China Acute Myocardial Infarction Registry Investigators. Impact of Marital Status on Management and Outcomes of Patients With Acute Myocardial Infarction: Insights From the China Acute Myocardial Infarction Registry. J Am Heart Assoc. 2022 Dec 6;11(23):e025671. doi: 10.1161/JAHA.122.025671. Epub 2022 Nov 29. PMID 36444834
- [Derived] Cui K, Fu R, Yang J, Xu H, Yin D, Song W, Wang H, Zhu C, Feng L, Wang Z, Wang Q, Lu Y, Dou K, Yang Y. Admission Blood Glucose and 2-Year Mortality After Acute Myocardial Infarction in Patients With Different Glucose Metabolism Status: A Prospective, Nationwide, and Multicenter Registry. Front Endocrinol (Lausanne). 2022 Jun 15;13:898384. doi: 10.3389/fendo.2022.898384. eCollection 2022. PMID 35784538
- [Derived] Cui K, Fu R, Yang J, Xu H, Yin D, Song W, Wang H, Zhu C, Feng L, Wang Z, Wang Q, Lu Y, Dou K, Yang Y; CAMI Registry Investigators. Stress hyperglycemia ratio and long-term mortality after acute myocardial infarction in patients with and without diabetes: A prospective, nationwide, and multicentre registry. Diabetes Metab Res Rev. 2022 Oct;38(7):e3562. doi: 10.1002/dmrr.3562. Epub 2022 Jul 13. PMID 35772392
- [Derived] Shi W, Ni L, Yang J, Fan X, Yu M, Yang H, Yu M, Yang Y; China Acute Myocardial Infarction (CAMI) Registry study group. The Clinical Impact of Proton Pump Inhibitors When Co-Administered With Dual Antiplatelet Therapy in Patients Having Acute Myocardial Infarction With Low Risk of Gastrointestinal Bleeding: Insights From the China Acute Myocardial Infarction Registry. Front Cardiovasc Med. 2021 Sep 22;8:685072. doi: 10.3389/fcvm.2021.685072. eCollection 2021. PMID 34631809
- [Derived] Shi W, Fan X, Yang J, Ni L, Su S, Yu M, Yang H, Yu M, Yang Y; China Acute Myocardial Infarction(CAMI) Registry Study Group. In-hospital gastrointestinal bleeding in patients with acute myocardial infarction: incidence, outcomes and risk factors analysis from China Acute Myocardial Infarction Registry. BMJ Open. 2021 Sep 7;11(9):e044117. doi: 10.1136/bmjopen-2020-044117. PMID 34493500
- [Derived] Song CX, Fu R, Yang JG, Xu HY, Gao XJ, Wang CY, Zheng Y, Jia SB, Dou KF, Yang YJ; CAMI Registry study group. Angiographic characteristics and in-hospital mortality among patients with ST-segment elevation myocardial infarction presenting without typical chest pain: an analysis of China Acute Myocardial Infarction registry. Chin Med J (Engl). 2019 Oct 5;132(19):2286-2291. doi: 10.1097/CM9.0000000000000432. PMID 31567475
- [Derived] Song C, Fu R, Li S, Yang J, Wang Y, Xu H, Gao X, Liu J, Liu Q, Wang C, Dou K, Yang Y. Simple risk score based on the China Acute Myocardial Infarction registry for predicting in-hospital mortality among patients with non-ST-segment elevation myocardial infarction: results of a prospective observational cohort study. BMJ Open. 2019 Sep 12;9(9):e030772. doi: 10.1136/bmjopen-2019-030772. PMID 31515430
- [Derived] Song C, Fu R, Dou K, Yang J, Xu H, Gao X, Wang H, Liu S, Fan X, Yang Y. Association between smoking and in-hospital mortality in patients with acute myocardial infarction: results from a prospective, multicentre, observational study in China. BMJ Open. 2019 Aug 30;9(8):e030252. doi: 10.1136/bmjopen-2019-030252. PMID 31471442
- [Derived] Leng W, Yang J, Fan X, Sun Y, Xu H, Gao X, Wang Y, Li W, Xu Y, Han Y, Jia S, Zheng Y, Yang Y; behalf CAMI Registry investigators. Contemporary invasive management and in-hospital outcomes of patients with non-ST-segment elevation myocardial infarction in China: Findings from China Acute Myocardial Infarction (CAMI) Registry. Am Heart J. 2019 Sep;215:1-11. doi: 10.1016/j.ahj.2019.05.015. Epub 2019 Jun 6. PMID 31255895
- [Derived] Fu R, Song CX, Dou KF, Yang JG, Xu HY, Gao XJ, Liu QQ, Xu H, Yang YJ. Differences in symptoms and pre-hospital delay among acute myocardial infarction patients according to ST-segment elevation on electrocardiogram: an analysis of China Acute Myocardial Infarction (CAMI) registry. Chin Med J (Engl). 2019 Mar 5;132(5):519-524. doi: 10.1097/CM9.0000000000000122. PMID 30807351
- [Derived] Dai Y, Yang J, Gao Z, Xu H, Sun Y, Wu Y, Gao X, Li W, Wang Y, Gao R, Yang Y; CAMI Registry study group. Atrial fibrillation in patients hospitalized with acute myocardial infarction: analysis of the china acute myocardial infarction (CAMI) registry. BMC Cardiovasc Disord. 2017 Jan 4;17(1):2. doi: 10.1186/s12872-016-0442-9. PMID 28052755
- [Derived] Sun H, Yang YJ, Xu HY, Yang JG, Gao XJ, Wu Y, Li W, Wang Y, Liu J, Jin C, Song L; CAMI Registry Study Group. [Survey of medical care resources of acute myocardial infarction in different regions and levels of hospitals in China]. Zhonghua Xin Xue Guan Bing Za Zhi. 2016 Jul 24;44(7):565-9. doi: 10.3760/cma.j.issn.0253-3758.2016.07.003. Chinese. PMID 27530939
- See also: China AMI registry — http://www.cami-r.com